CLINICAL TRIAL: NCT07241637
Title: The Effect of Tele-Yoga Application on Chronic Pelvic Pain, Fatigue and Quality Of Life In Women With Endometriosis Diagnosis
Brief Title: Effect of Tele-Yoga on Pain, Fatigue, and Quality of Life in Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Melek Hava Köprülü, PhD Student, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AnkaraU-HEM-RK-02
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Pain; Endometriosis
Keywords: Pelvic Pain; Yoga; Fatigue; Quality of Life; Endometriosis
MeSH Terms: conditions — Pelvic Pain; Endometriosis; Fatigue

STUDY DESIGN:
Intervention Model Description: A comprasion of the two groups to be assigned as experimental and control groups will be made.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Group (Experimental): The researcher will conduct online Tele-yoga sessions with patients diagnosed with endometriosis and experiencing pain in the intervention group using a computer or tablet. The program will include a total of 16 individual sessions, held twice a week for eight weeks, each lasting 60 minutes. Sessions will be conducted live via the Google Meet platform between the researcher and the participant. The schedule for the following week will be determined after the second session each week. All sessions will take place in a private setting chosen by the participant, ensuring privacy and comfort, and no screenshots or video recordings will be taken during the sessions.The intervention will begin with breathing exercises and a 10-minute meditation in the Sukhasana pose, followed by a 10-minute warm-up of stretching and mobilization. Then, a 35-minute yoga flow combining various asanas with breathing techniques will be performed, ending with 5 minutes of deep relaxation in the Savasana pose
  Interventions: Behavioral: Tele-Yoga Group
- Control Group (No Intervention): No intervention will be applied to the control group. Participants will be followed for eight weeks, and they will be expected to complete the scales at the end of the eighth week

INTERVENTIONS:
Behavioral: Tele-Yoga Group — Tele-yoga is a telerehabilitation method that enables the delivery of yoga-based rehabilitation services through electronic systems. Initially developed for emergency management, this approach has become effective in daily practice with the increasing cost of treatment and the privatization of healthcare services. Yoga is a practice that can be adapted to the individual needs of each woman. In women with endometriosis, yoga helps develop a different response to pain through mindful attention to painful areas, relaxation postures, breathing techniques, and movement sequences
  Arms: Tele-Yoga Group

SUMMARY:
This study aims to examine the effects of Tele-yoga on chronic pelvic pain, fatigue, and quality of life in patients diagnosed with endometriosis. It will be conducted as a single-center, randomized controlled experimental study design.

DETAILED DESCRIPTION:
Endometriosis is a chronic, estrogen-dependent condition affecting approximately 10% of women of reproductive age worldwide. In Türkiye, it is estimated that around 2.4 million women are diagnosed with endometriosis. The disease is commonly associated with symptoms such as chronic pelvic pain (CPP), dysmenorrhea, dyspareunia, and infertility, among which CPP is the most prevalent. Endometriosis-related pain is typically recurrent and progressive, significantly impairing women's daily activities and overall quality of life.

Fatigue is another frequently reported symptom among women with endometriosis. Evidence indicates that fatigue is substantially more common in this population compared to the general female population and has a detrimental impact on both physical and psychological well-being. The coexistence of chronic pain and fatigue further exacerbates the negative effects of endometriosis on quality of life.

In recent years, there has been growing interest in Complementary and Integrative Health Approaches (CIHA) for managing pain and fatigue associated with endometriosis. The National Institute for Health and Care Excellence (NICE) guidelines emphasize the importance of multidisciplinary and mind-body-based strategies in endometriosis management. Yoga, recognized by the World Health Organization (WHO) as a complementary health practice, integrates physical postures, breathing exercises, and meditation. It is a low-cost, non-invasive intervention known to promote relaxation and reduce pain, stress, and fatigue.

Telerehabilitation enables the remote delivery of such interventions through digital technologies, improving accessibility and continuity of care. However, there is a limited number of studies investigating telerehabilitation-based yoga interventions among women experiencing chronic pelvic pain due to endometriosis.

Therefore, this project aims to examine the effects of Tele-yoga on chronic pelvic pain, fatigue, and quality of life in women diagnosed with endometriosis. The findings of this research are expected to contribute to developing holistic, accessible, and evidence-based management strategies for women living with endometriosis

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the research
* Able to communicate effectively and have no language barriers
* Have at least a primary school education
* Are 18 years of age or older and premenopausal
* Are not pregnant
* Have no health problems that would prevent them from practicing yoga
* Do not exercise regularly / do not exercise more than three times per week
* Have not received physical therapy within the past three months
* Have not undergone any pelvic surgery within the past year
* Do not have surgical treatment planned for endometriosis
* Do not have any other injury or disease causing pelvic pain
* Have mild (1-3) or moderate (4-6) chronic pelvic pain
* Have access to a computer, phone, or tablet with a camera and an available internet connection to participate in online sessions

Exclusion Criteria:

* Those who wish to withdraw at any stage of the research
* Those who do not attend all Tele-yoga sessions
* Those who begin regular exercise or physical therapy during the study period
* Those who become pregnant during the study
* Those who use any Complementary or Alternative Medicine (CAM) method during the intervention
* Those who undergo surgical treatment during the course of the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | The scale will be administered to all groups before the intervention begins and after the intervention is completed (at the end of the eighth week)
  In patients diagnosed with endometriosis, the Numerical Rating Scale (NRS) is used to assess pain intensity by having the patient rate their perceived pain on a scale from 0 to 10.A value of 0 is considered "no pain," while a value of 10 is considered "the worst pain imaginable." Patients are asked to circle the number representing the amount of pain they experience during the assessment. As the number on the scale increases, the pain increases.

SECONDARY OUTCOMES:
The Fatigue Severity Scale (FSS) | The scale will be administered to all groups before the intervention begins and after the intervention is completed (at the end of the eighth week).
  The Fatigue Severity Scale (FSS) is used to determine how fatigued the patient has felt over the past week, including the day the test is administered.
The Endometriosis Health Profile-5 (EHP-5) | The scale will be administered to all groups before the intervention begins and after the intervention is completed (at the end of the eighth week)
  The Endometriosis Health Profile-5 (EHP-5) is used to assess the impact of endometriosis on women's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Özdemir, Principal Investigator — Ankara University
Locations (1):
- Ankara University Nursing Faculty, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No